CLINICAL TRIAL: NCT04500210
Title: A Double-blind, Randomized, Parallel Group, Phase III Comparative Study of Turmeric Extract and Placebo to Patients With Mild to Moderate Arthrosis of the Knee and or Hip.
Brief Title: Comparative Study of Turmeric Extract in Patients With Arthrosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaj Winther Hansen (Other)
Responsible Party: Sponsor-Investigator, Kaj Winther Hansen, professor, MD, DMsCi, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tr-01
Record Dates: First submitted 2020-01-03; First posted 2020-08-05 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2020-07

CONDITIONS: Arthralgia; Stiffness of Unspecified Joint, Not Elsewhere Classified; Disturbance of Activity and Attention; Quality of Life
Keywords: Arthralgia, stiffness of joints, quality of life
MeSH Terms: conditions — Arthralgia | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Half of the volunteers are given placebo and half of the volunteers are given Turmeric extract
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): one capsule daily
  Interventions: Dietary Supplement: Placebo
- Turmeric extract (Active Comparator): one capsule daily
  Interventions: Dietary Supplement: Turmeric

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo in gelatin capsules
  Arms: Placebo
Dietary Supplement: Turmeric — Turmeric in gelatin capsules
  Arms: Turmeric extract

SUMMARY:
The aim of this study is to test if an extract of Turmeric can alleviate symptoms of osteoarthritis in volunteers with osteoarthritis of the hip and or knee.

DETAILED DESCRIPTION:
The included volunteers, who are devided into two groups either placebo or turmeric extract, will be tested using WOMAC questionnaires focussing on pain, stiffness and daily activity. In addition different aspects of quality of life will be evaluated and the consumption of rescue medication will be recorded in patients personal diary.

The treatment period is 3 month with the posibility to continue for an additional 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* 40 years of age or more
* Osteoarthritis of the hip and or the knee
* Suffering from pain in the hip and or knee -

Exclusion Criteria:

* If volunteers are on a waiting list for hip or knee surgery
* If the volunteers are involved in an other clinical trial
* If the volunteers are taking other herbal remedies, which canhav influende on # Osteoarthritis.
* Abusers of alcohol and drugs
* Volunteers not easy to cope with

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Pain | 3 month
  Difference in WOMAC pain on a 100 mm VAS scale (high levels worse)
Pain | 6 month
  Difference in WOMAC pain on a 100 mm VAS scale (high levels worse)
ADL (Activity of daily living) | 3 month
  Difference in WOMAC ADL on a 100 mm VAS scale (high levels worse)
ADL (Activity of daily living) | 6 month
  Difference in WOMAC ADL on a 100 mm VAS scale (high levels worse)
Rescue medication | 3 month
  Consumption of rescue medication from diaries (mg)
Rescue medication | 6 month
  Consumption of rescue medication from diaries (mg)

SECONDARY OUTCOMES:
Stiffness of joints | 3 month
  Difference in stiffness of joints on a 100 mm VAS scale (higher values worse)
Stiffness of joints | 6 month
  Difference in stiffness of joints on a 100 mm VAS scale (higher values worse)
The volunteer evaluation of Global Disease Severity (PGAD) | 3 month
  PGAD is measured on a 100 mm VAS scale (higher values worse)
The volunteer evaluation of Global Disease Severity (PGAD) | 6 month
  PGAD is measured on a 100 mm VAS scale (higher values worse)

OTHER OUTCOMES:
SF-12 (Quality of life) | 3 month
  Quality of life estimated on a numerical scale (1-3 and 1-6)
SF-12 (quality of life) | 6 month
  Quality of life estimated on a numerical scale (1-3 and 1-6)

CONTACTS AND LOCATIONS:
Overall Officials: Kaj W Hansen, Prof, DMSCi, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark